CLINICAL TRIAL: NCT03034161
Title: Thermal Imaging to Identify Distinct Temperature Patterns in Various Stages of Pressure Ulcers
Status: Withdrawn | Type: Observational
Why Stopped: lack of funding
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Other Study IDs: 206042
Record Dates: First submitted 2017-01-25; First posted 2017-01-27 (Estimated); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Decubitus Ulcer; Pressure Ulcer
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Stage I Pressure Ulcer: Ten patients with a Stage I decubitus pressure ulcer will be included to be analyzed with a thermal imaging camera.
  Interventions: Device: Thermal imaging
- Stage II Pressure Ulcer: Ten patients with a Stage II decubitus pressure ulcer will be included to be analyzed with a thermal imaging camera.
  Interventions: Device: Thermal imaging
- Stage III Pressure Ulcer: Ten patients with a Stage III decubitus pressure ulcer will be included to be analyzed with a thermal imaging camera.
  Interventions: Device: Thermal imaging
- Stage IV Pressure Ulcer: Ten patients with a Stage IV decubitus pressure ulcer will be included to be analyzed with a thermal imaging camera.
  Interventions: Device: Thermal imaging

INTERVENTIONS:
Device: Thermal imaging — Thermal imaging of the various stages of pressure ulcer will be analyzed to determine if a recognizable pattern of thermal distribution can be identified which can then be applied to identify patients at risk of developing pressure ulcers at an earlier stage in their hospital course.

SUMMARY:
40 patients total with pressure ulcers with a decubitus pressure ulcer will be included in this study. Ten patients with a Stage I, II, III, and IV decubitus pressure ulcer will be included to be analyzed with a thermal imaging camera. Thermal imaging of the various stages of pressure ulcer will be analyzed to determine if a recognizable pattern of thermal distribution can be identified which can then be applied to identify patients at risk of developing pressure ulcers at an earlier stage in their hospital course.

DETAILED DESCRIPTION:
This study will be a single-center prospective Phase I study in which the use of a thermal imaging camera will be used to obtain imaging data on decubitus ulcers of various stages. The data collected during this study will be used to determine if stage-specific thermal distribution patterns can be identified. This information will then be used to design future studies in which patients are risk for the development of pressure ulcers are screened for the presence of pressure ulcers not detectable upon physical examination so that preventative measures and treatments can be instituted.

A total of 40 patients with pressure decubitus ulcers will be recruited for inclusion in this study. The investigators plan to enroll ten patients with each stage of pressure ulcer (i.e. Stage I-IV), which will provide the investigators with a set of thermal imaging data from which the investigators will determine if thermal distribution patterns unique to each stage of pressure ulcer can be identified. It is anticipated that 40 patients who meet the inclusion criteria and distribution of pressure ulcer staging will be enrolled within one year of the start date of this study.

The investigators are planning a study of a continuous response variable from independent control and experimental subjects with 1 control(s) per experimental subject. It is estimated that the response within each subject group will be normally distributed with standard deviation 25. If the true difference in the experimental and control means is 35, the investigators will need to study 9 experimental subjects and 9 control subjects to be able to reject the null hypothesis that the population means of the experimental and control groups are equal with probability (power) 0.8. The Type I error probability associated with this test of this null hypothesis is 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients with sacral/heel pressure ulcers, admitted to University of Arkansas for Medical Sciences (UAMS) inpatient services.
* Patients 18-years old or older.
* Patients have an expected survival of > 48 hours

Exclusion Criteria:

* Patients not compliant with obtaining thermal imaging.
* Patients not expected to survive for 48 hours.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with sacral/heel pressure ulcers
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-04-29 (Actual); Study Completion 2019-04-29 (Estimated)

PRIMARY OUTCOMES:
Difference in temperature between a Stage I, Stage 2, Stage 3 and Stage 4 decubitus pressure ulcer as measured by using the thermal imaging camera. | Up to one year
  Each subject will receive one temperature measurement during inpatient status of the decubitus pressure ulcer using the thermal imaging camera.

CONTACTS AND LOCATIONS:
Overall Officials: Jacob T Carlson, MD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: Undecided